CLINICAL TRIAL: NCT04594590
Title: A Natural History Study of Neurodegeneration and Optic Atrophy Caused by SLC25A46 Mutations in Pediatric and Adult Patients
Brief Title: Natural History Study of SLC25A46 Mutation-related Mitochondriopathy
Status: Completed | Type: Observational
Sponsor: State University of New York at Buffalo (Other)
Collaborators: Hadley Jo Foundation (Unknown)
Responsible Party: Principal Investigator, Taosheng Huang, Principal Investigator, State University of New York at Buffalo
Other Study IDs: STUDY00004513-SLC
Record Dates: First submitted 2020-10-13; First posted 2020-10-20 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Neurodegenerative Disease, Hereditary; Mitochondrial Diseases; Optic Atrophy
Keywords: Neurodegeneration; Mitochondrial disease; Optic atrophy; SLC25A46; Mitochondrial fission
MeSH Terms: conditions — Heredodegenerative Disorders, Nervous System; Mitochondrial Diseases; Optic Atrophy; Nerve Degeneration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — The medical records will be retained for all patients. For select patients, blood, DNA, skin punch biopsies will also be obtained for the purpose of genetic and biochemical analysis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with SLC25A46 deficiency: Male and female patients from age 2 to age 65 with clinically confirmed SLC25A46 mutations. Both living and deceased patients will be included, if eligible. For deceased patients, the patient's medical history records will be reviewed, and an interview of the parent(s) or caregiver(s) will be performed.
  Interventions: Genetic: Mutation analysis

INTERVENTIONS:
Genetic: Mutation analysis — The investigators will sequence DNA samples from the patients or their families.

SUMMARY:
The purpose of the study is to systematically characterize the clinical course of the progressive neuropathy and optic atrophy observe in pediatric and adult patients with biallelic mutations in the solute carrier family 25 member 46 (SLC25A46) gene.

DETAILED DESCRIPTION:
The number of mitochondria in the cell is dynamic and is regulated by two opposite processes, namely fission and fusion. Proteins in both the inner mitochondrial membrane (IMM) and the outer mitochondrial membrane (OMM) are involved in mediating these two processes, including OPA1, MFN2 and SLC25A46. Recent work by the investigators as well as other research groups has shown that mutations in SLC25A46 cause abnormal mitochondrial fusion, leading to optic nerve atrophy, axonal peripheral neuropathy and cerebellar degeneration by interfering with mitochondrial fission. Recently, the investigators have used CRISPR genome editing to generate a global Slc25a46 KO mouse model with complete loss of SLC25A46 in all tissues (PMID: 28934388). Similar to patients with biallelic mutations in SLC25A46, these mice exhibit severe ataxia, optic atrophy, peripheral neuropathy related to axonal degeneration, and demyelination due to mitochondrial hyperfusion and defective energy production. In these mice, histological staining revealed a hypotrophic cerebellum with a severe loss of Purkinje cells (PCs) and/or stunted PC dendrites while electron microscopy revealed enlarged mitochondria with swollen cristae and other abnormal morphologies in PC dendrites and sciatic nerves. Furthermore, in primary culture, PCs from these mice exhibited abnormal mitochondrial distribution and movement.

These findings provide compelling evidence indicating that SLC25A46 plays an important role in the regulation of mitochondrial dynamics-including fusion/fission, distribution, and movement, as well as the maintenance of cristae architecture-and that loss of SLC25A46 function has a particularly severe effect on a distinct subset of neuron types with long axonal processes. More recently, the investigators have shown that AAV-based gene therapy can produce dramatic improvements in their Slc25a46 mutant mouse model (PMID: 31943007). These studies in the Slc25a46 mouse model provide the foundation for uncovering the mechanism whereby these this gene causes disease in humans, as well as lay the groundwork for the possible use of gene therapy to ameliorate the disease phenotype in patients.

However, despite this progress, there remains only a handful of studies published on Slc25a46 and the consequences of loss of Slc25a46 function in humans. Given that human SLC25A46-associated phenotypes overlap substantially with DOA and CMT2A, further study of this rare condition presents an opportunity not only to better understand and treat SLC25A46-related disease, but also to elucidate the broader mechanistic link between neurodegeneration and abnormal mitochondrial dynamics. Thus, in order to better understand the clinical manifestations of SLC25A46-related disease and to help lay the groundwork for eventual clinical trials of gene therapy or drug-based treatments, the investigators propose this natural history study of pediatric as well as adult patients with biallelic mutations in the SLC25A46 gene.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are clinically diagnosed with biallelic mutations in the SLC25A46 gene
* Male and female patients from 2 to 65 years of age
* Patients who have consented to the study
* In the case of a deceased patient whose parent(s) and/or legal guardian(s) have provided informed consent for study participation, the investigators will review the patient's medical records to determine study eligibility.

Exclusion Criteria:

* Significant postnatal complications or congenital anomalies that are not known to be associated with SLC25A46 dysfunction
* Patient has received any experimental treatment for SLC25A46 dysfunction within the 6 months prior to enrollment, or is expected to receive any such therapy during the study period

Ages: 0 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2020-11-03 (Actual); Primary Completion 2023-08-17 (Actual); Study Completion 2023-08-17 (Actual)

PRIMARY OUTCOMES:
Custom Medical History Questionnaire for Patients with SLC25A46 Mutation-related Mitochondriopathy | 3 years
  In addition to a standard medical history, patients or their legal guardians will be asked to complete a custom medical history questionnaire tailored toward conditions commonly observed in patients with biallelic SLC25A46 mutations. The items that will be asked about in this questionnaire are as follows:
  1. Known mutations in SLC25A46
  2. Any family history of illness
  3. Complications of pregnancy
  4. Premature birth
  5. Complications with birth
  6. Developmental delay
  7. Developmental regression
  8. Abnormal size of brain
  9. Movement disorders (ataxia, dystonia, etc.)
  10. Seizures
  11. Optic atrophy in eye exam
  12. Vision loss
  13. Other vision problems (color, eye movement)
  14. Hypotonia (muscle weakness or lack of tone)
  15. Electromyogram (EMG)
  16. Muscle biopsy
  17. Spasticity (muscle stiffness or tightness)
  18. Brain MRI performed?
  19. Electroencephalogram (EEG)
Retrospective examination of the medical records of patients with SLC25A46 Mutation-related Mitochondriopathy | 3 years
  With the informed consent of the patients or their parent(s) and/or legal guardian(s), the investigators will perform a retrospective examination of the medical records of both living and deceased patients with confirmed biallelic SLC25A46 mutations.
Eye assessments to evaluate ocular health | 3 years
  Visual acuity examination will be performed to determine the patient's clarity or sharpness of vision.
Growth and development (height) | 3 years
  World Health Organization (WHO) growth charts will be used to document height in centimeters (cm) for patients ranging from ages 5 to 19 years old. Routine methods will be used to document height for all other age groups.
Growth and development (weight) | 3 years
  World Health Organization (WHO) growth charts will be used to document weight in kilograms (kg) for pediatric patients age 5 to 10 years old. Routine methods will be used to document weight for all other age groups.
Growth and development (BMI) | 3 years
  World Health Organization (WHO) growth charts will be used to document Body Mass Index (BMI) in kilograms per meter square for patients age 5 to 19 years old. Routine methods will be used to document BMI for all other age groups.

CONTACTS AND LOCATIONS:
Overall Officials: Taosheng Huang, Principal Investigator — State University of New York at Buffalo
Locations (1):
- UBMD Pediatrics, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abrams AJ, Hufnagel RB, Rebelo A, Zanna C, Patel N, Gonzalez MA, Campeanu IJ, Griffin LB, Groenewald S, Strickland AV, Tao F, Speziani F, Abreu L, Schule R, Caporali L, La Morgia C, Maresca A, Liguori R, Lodi R, Ahmed ZM, Sund KL, Wang X, Krueger LA, Peng Y, Prada CE, Prows CA, Schorry EK, Antonellis A, Zimmerman HH, Abdul-Rahman OA, Yang Y, Downes SM, Prince J, Fontanesi F, Barrientos A, Nemeth AH, Carelli V, Huang T, Zuchner S, Dallman JE. Mutations in SLC25A46, encoding a UGO1-like protein, cause an optic atrophy spectrum disorder. Nat Genet. 2015 Aug;47(8):926-32. doi: 10.1038/ng.3354. Epub 2015 Jul 13. PMID 26168012
- [Background] Li Z, Peng Y, Hufnagel RB, Hu YC, Zhao C, Queme LF, Khuchua Z, Driver AM, Dong F, Lu QR, Lindquist DM, Jankowski MP, Stottmann RW, Kao WWY, Huang T. Loss of SLC25A46 causes neurodegeneration by affecting mitochondrial dynamics and energy production in mice. Hum Mol Genet. 2017 Oct 1;26(19):3776-3791. doi: 10.1093/hmg/ddx262. PMID 28934388
- [Background] Yang L, Slone J, Li Z, Lou X, Hu YC, Queme LF, Jankowski MP, Huang T. Systemic administration of AAV-Slc25a46 mitigates mitochondrial neuropathy in Slc25a46-/- mice. Hum Mol Genet. 2020 Mar 13;29(4):649-661. doi: 10.1093/hmg/ddz277. PMID 31943007
- [Background] Qiu K, Zou W, Fang H, Hao M, Mehta K, Tian Z, Guan JL, Zhang K, Huang T, Diao J. Light-activated mitochondrial fission through optogenetic control of mitochondria-lysosome contacts. Nat Commun. 2022 Jul 25;13(1):4303. doi: 10.1038/s41467-022-31970-5. PMID 35879298
- [Background] Zou W, Chen Q, Slone J, Yang L, Lou X, Diao J, Huang T. Nanoscopic quantification of sub-mitochondrial morphology, mitophagy and mitochondrial dynamics in living cells derived from patients with mitochondrial diseases. J Nanobiotechnology. 2021 May 13;19(1):136. doi: 10.1186/s12951-021-00882-9. PMID 33985528
- See also: Link to the official website for the "Hadley Jo Foundation" — https://hadleyjofoundation.org/